CLINICAL TRIAL: NCT04632667
Title: CATCH Healthy Smiles: A Cluster-RCT of an Elementary School Oral Health Intervention
Brief Title: CATCH Healthy Smiles:An Elementary School Oral Health Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SPH-19-0838
Record Dates: First submitted 2020-10-12; First posted 2020-11-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Schools will be cluster randomized to the intervention or comparison group
Who Masked: Investigator
Masking Description: For post measurements, all data collection staff will be blinded to the intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparison School Group (Active Comparator)
  Interventions: Behavioral: Comparison School Group
- Intervention School Group (Experimental)
  Interventions: Behavioral: Intervention School Group

INTERVENTIONS:
Behavioral: Comparison School Group — All control schools will receive training and materials for the CATCH sun safety curriculum. Ray and the Sunbeatables®: A Sun Safety Curriculum is an evidence-based curriculum educates children, parents and teachers about sun protection and promotes sun safety behaviors in an effort to reduce children's lifetime risk of developing skin cancer. Training will be conducted with booster trainings yearly.
  Arms: Comparison School Group
Behavioral: Intervention School Group — This intervention includes toothbrushing which will be implemented as a daily activity to develop skills and technique,classroom curriculum, which includes theory-based interactive lessons on oral health care,the physical education component consisting of an activity box containing different structured physical activities that will integrate the nutrition and oral health education messages, all cafeteria-based intervention materials including the "tooth friendly" Eat Smart guide, signage, nutrition labeling, menu planning and labeling using the tooth-friendly Go-Slow-Whoa CATCH terminology will be provided to the food service staff that is displayed across the cafeteria and sent home to parents and parents will be provided with tools and tips for maintaining oral health with website resources,parent-child homework activities, send-home infographics on dental care, parent-monitored tracking of child oral health,family fun nights in schools, and social media.
  Arms: Intervention School Group

SUMMARY:
The purpose of this study is to clinically evaluate the effects of a school-based behavioral intervention, CATCH Healthy Smiles, to reduce the risk of dental caries in a cohort of kindergarten through 2nd grade (K-2) children serving low-income, ethnically-diverse children,to determine the impact of CATCH Healthy Smiles on child behavioral, psychosocial, and environmental outcomes beginning in K through 2nd grade, compared to children in the control schools and to examine the extent to which the child behavioral, psychosocial, and environmental factors mediate the improvements in child caries risk.

ELIGIBILITY:
Inclusion Criteria:

For schools:

* greater than 75% of the children enrolled in the dree/reduced school lunch program.
* enrolling children in grade K in the 2021-2022 school year.
* agree to implement the CATCH Healthy Smiles program and agreed to participate in the measurements

For parent and child to participate in the measures:

* ability of the parent to speak and read in English or Spanish at the 4th grade level,
* child enrolled in the participating school in grade K in the 2021-2022 school year
* child ability to participate in the regular activities at the school

Exclusion Criteria:

-No congenital dental conditions such as cleft palate, children with enamel hypoplasia, severe fluorosis, or special dental setting needs.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1084 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of tooth and tooth surfaces that became decayed or were treated for dental caries (by filling or extraction) | Baseline(beginning of kindergarten)
Number of tooth and tooth surfaces that became decayed or were treated for dental caries (by filling or extraction) | end of year 1(Kindergarten)
Number of tooth and tooth surfaces that became decayed or were treated for dental caries (by filling or extraction) | end of year 2(first grade)
number of tooth and tooth surfaces that became decayed or were treated for dental caries (by filling or extraction) | end of year 3( second grade)

SECONDARY OUTCOMES:
Number of children with good oral hygiene as measured by the child plaque index | Baseline
  The plaque score will be measured using the plaque index of Silness and Loe. Six teeth will be examined for presence of plaque/ materia alba and food remnants and calculus. The index will be a numerical score (0-3) as follows: 0 = No Debris or stain; 1 = Soft debris or stain covering no more than 1/3 of tooth surface; 2 = Soft debris or stain covering more than 1/3 of tooth surface and less than 2/3 of tooth surface; 3 = Soft debris or stain covering more than 2/3 of tooth surface.
Number of children with good oral hygiene as measured by the child plaque index | end of year 1 about 9 months form start of intervention
  The plaque score will be measured using the plaque index of Silness and Loe. Six teeth will be examined for presence of plaque/ materia alba and food remnants and calculus. The index will be a numerical score (0-3) as follows: 0 = No Debris or stain; 1 = Soft debris or stain covering no more than 1/3 of tooth surface; 2 = Soft debris or stain covering more than 1/3 of tooth surface and less than 2/3 of tooth surface; 3 = Soft debris or stain covering more than 2/3 of tooth surface.
Number of children with good oral hygiene as measured by the child plaque index | end of year 2 about 23 months from start of intervention
  The plaque score will be measured using the plaque index of Silness and Loe. Six teeth will be examined for presence of plaque/ materia alba and food remnants and calculus. The index will be a numerical score (0-3) as follows: 0 = No Debris or stain; 1 = Soft debris or stain covering no more than 1/3 of tooth surface; 2 = Soft debris or stain covering more than 1/3 of tooth surface and less than 2/3 of tooth surface; 3 = Soft debris or stain covering more than 2/3 of tooth surface.
Number of children with good oral hygiene as measured by the child plaque index | end of year 3 about 33 months form start of intervention
  The plaque score will be measured using the plaque index of Silness and Loe. Six teeth will be examined for presence of plaque/ materia alba and food remnants and calculus. The index will be a numerical score (0-3) as follows: 0 = No Debris or stain; 1 = Soft debris or stain covering no more than 1/3 of tooth surface; 2 = Soft debris or stain covering more than 1/3 of tooth surface and less than 2/3 of tooth surface; 3 = Soft debris or stain covering more than 2/3 of tooth surface.
Child dietary intake as measured by the Block food frequency screener | Baseline
  This tools helps to find out how many times a week different kinds of food was consumed and how much quantity of food was consumed each day
Child dietary intake as measured by the Block food frequency screener | end of year 1
  This tools helps to find out how many times a week different kinds of food was consumed and how much quantity of food was consumed each day
Child dietary intake as measured by the Block food frequency screener | end of year 2
  This tools helps to find out how many times a week different kinds of food was consumed and how much quantity of food was consumed each day
Child dietary intake as measured by the Block food frequency screener | end of year 3
  This tools helps to find out how many times a week different kinds of food was consumed and how much quantity of food was consumed each day
Child and parent behavioral, psychosocial and environmental factors will be measured using self-report surveys | Baseline
Child and parent behavioral, psychosocial and environmental factors will be measured using self-report surveys | end of year 1 about 9 months from start of intervention
Child and parent behavioral, psychosocial and environmental factors will be measured using self-report surveys | End of year 2 about 23 months from start of intervention
Child and parent behavioral, psychosocial and environmental factors will be measured using self-report surveys | End of year 3 about 33 months from start of intervention
Number of times a child brushes their teeth a day | Baseline
Number of times a child brushes their teeth a day | end of year 1 about 9 months from start of intervention
Number of times a child brushes their teeth a day | End of year 2 about 23 months from start of intervention
Number of times a child brushes their teeth a day | End of year 3 about 33 months from start of intervention
Change in Body Mass Index (BMI) | baseline, end of Year 1, Year 2 and Year 3
  Child height and weight measured at the school using stadiometers and digital scales respectively.
Change in Child Oral health quality of life measured using parent self-report surveys | baseline, end of Year 1, Year 2 and Year 3
Frequency of flossing teeth for the child measured using parent self-report surveys | Baseline
Frequency of flossing teeth for the child measured using parent self-report surveys | end of year 1
Frequency of flossing teeth for the child measured using parent self-report surveys | end of year 2
Frequency of flossing teeth for the child measured using parent self-report surveys | end of year 3

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuang RJ, Byrd-Williams C, Yamal JM, Johnson K, Kelder S, Nelson S, Mofleh D, Sharma SV. Design for a cluster randomized controlled trial to evaluate the effects of the CATCH Healthy Smiles school-based oral health promotion intervention among elementary school children. Contemp Clin Trials Commun. 2022 Nov 5;30:101033. doi: 10.1016/j.conctc.2022.101033. eCollection 2022 Dec. PMID 36387989